CLINICAL TRIAL: NCT04129593
Title: Self Awakening and Snoozing Effects on the Cortisol Awakening Response
Acronym: SASECAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Notre Dame (Other)
Responsible Party: Principal Investigator, Stephen Mattingly, Post-Doctoral Reserarcher, University of Notre Dame
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19-08-5534
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Cortisol Awakening Response

STUDY DESIGN:
Intervention Model Description: Participants will undergo 1 of 2 conditions on Saturday and Sunday; Self awakening and natural waking, or snooze and natural waking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self Awakening (Experimental): Participant will intend to wake up at a specific time before going to bed.
  Interventions: Behavioral: Self Awakening - Natural Waking
- Snooze (Experimental): Participant will set multiple alarms before bed to wake at a specific time.
  Interventions: Behavioral: Snooze - Natural waking

INTERVENTIONS:
Behavioral: Self Awakening - Natural Waking — subjects in this arm will be assigned to natural waking and self awaking conditions on Saturday and Sunday. they will be counterbalanced equally between Saturday: natural waking, Sunday: self awakening and Saturday: self awakening, Sunday: natural waking.
  Arms: Self Awakening
Behavioral: Snooze - Natural waking — subjects in this arm will be assigned to snooze and natural waking conditions on Saturday and Sunday. they will be counterbalanced equally between Saturday: snooze, Sunday: natural waking and Saturday: natural waking, Sunday: snooze.
  Arms: Snooze

SUMMARY:
One third of American adults and teens are sleep deprived, and less than 8% of highschool students achieve recommended amounts of sleep. 85% of Americans consume caffeine daily, and a pilot study we conducted suggests over half of working professionals snooze. Sleep deprivation results in sleep inertia (grogginess) upon waking, and many behaviors are employed to reduce the negative effects of sleep inertia, including self-awakening (SA - going to bed intending to wake at a specific time) and snoozing (setting multiple alarms or using a snooze function). SA reduces sleep inertia and may increase stress system activity before waking, but snoozing is virtually unstudied, though alarms can also increase stress system activity. The cortisol awakening response (CAR) is a boost in the stress hormone, cortisol, that occurs naturally upon waking. The CAR is thought to reduce sleep inertia and to prepare for the anticipated stressors of the day, and this physiological process can be blunted in those who are sleep deprived and/or have medical or psychiatric conditions. This proposal seeks to increase the CAR in healthy individuals through SA and snooze interventions. Participants receive a commercial wearable at the beginning of the week that tracks sleep and heart rate, as well as a study phone that monitors the sleep environment, tracks alarms, and administers cognitive tests after waking to determine sleep inertia. These devices allow a development of baseline waking behavior. On Saturday and Sunday mornings undergo additional including a higher quality heart rate monitor and body temperature sensor. Participants also undergo 2 of 3 conditions; SA, snoozing, and natural waking. In the SA condition, participants intend to wake up 7 hours after they go to bed. In the snooze condition, participants set multiple alarms to terminate 7 hours after bedtime. In the natural waking condition, participants wake up normally. Upon waking, participants provide multiple saliva samples and undergo cognitive performance assessments and answer questions about mood for 1 hour. By comparing the cortisol samples between conditions, we can determine if SA and/or snoozing increases the CAR relative to natural waking. The cognitive performance tests will also be tested between conditions to determine if the interventions reduce sleep inertia and/or increase stress system activity. Interventions that specifically increase the CAR and reduce sleep inertia in healthy individuals could then be tested for those who have blunted CAR, e.g. chronic pain sufferers, to improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

Legally able to provide consent -

Exclusion Criteria:

Not legally able to provide consent

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Cortisol Awakening Response | 4 samples: immediately upon waking, 15 minutes post waking, 30 minutes post waking, and 45 minutes post waking. Samples are provided for 10 minutes.
  A biomarker for Hypothalamic Pituitary Adrenal activity; a naturally occurring increase in cortisol upon waking.

SECONDARY OUTCOMES:
Heart Rate upon waking | Heart rate will be continuously assessed for the entire week. Note: data is divided into 1 minute bin averages.
  Stress activity before waking can increase heart rate. We want to see if alarms and / or snoozing increase heart rate upon waking
Sleep inertia - cognitive throughput | During weekdays, sleep inertia will be assessed immediately upon waking, duration is 5 minutes. On Saturday and Sunday, they will be assessed at wake + 10 minutes, wake +25 minutes, wake + 40 minutes, and wake + 55minutes.
  sleep inertia is a marked decrease in cognitive abilities upon waking. We wish to see if cognitive performance upon waking is better when snoozing or self awakening.

IPD SHARING:
Plan to Share IPD: No